CLINICAL TRIAL: NCT02148471
Title: Non-alcoholic Steatohepatitis Versus Simple Hepatic Steatosis: Is There a Difference in the Nutritional Factors Influencing Lipid Perioxidation and Inflammation?
Brief Title: Fatty Acids, Genes and Microbiota in Fatty Liver
Status: Completed | Type: Observational
Sponsor: Johane Allard (Other)
Collaborators: Canadian Liver Foundation (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); American College of Gastroenterology (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Prof. Dr., University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 03-0505-A
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Nonalcoholic Fatty Liver Disease; Steatosis; Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic fatty liver disease; Steatosis; Nonalcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA - samples retained, with potential for extraction of DNA from at least one of the types of samples retained (e.g., frozen tissue, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: Healthy living liver donors with healthy liver on imaging and/or liver histology
- Simple steatosis: Patients with non-alcoholic fatty liver disease confirmed by liver biopsy with a diagnosis of simple steatosis
- Nonalcoholic steatohepatitis: Patients with non-alcoholic fatty liver disease confirmed by liver biopsy with a diagnosis of steatohepatitis
- Minimal findings: Patients undergoing liver biopsy because of suspected fatty liver but nonspecific findings on liver histology. This group was initially used as a control group. Later in the study, this group was replaced by healthy donors as true healthy controls.

SUMMARY:
The first aim of this study is to assess oxidative stress and nutritional status in patients with elevated liver enzymes who were found to have either simple steatosis (SS) or nonalcoholic steatohepatitis (NASH) or normal histological findings on liver biopsy by measuring liver lipid peroxides and tumor necrosis factor (TNF)-α, liver pathology and immunohistochemistry, liver function tests, liver and red blood cell membrane fatty composition, insulin resistance (IR) parameters, plasma lipid peroxides, plasma antioxidant vitamins and antioxidant power, lipid profile, subject demographics, medical history and medication use. The second aim is to detect differences in hepatic gene expression (messenger RNA, mRNA) and epigenetic regulation (micro RNA, miRNA) between patients with SS or NASH and healthy controls, in addition to determine in patients with non-alcoholic fatty liver disease (NAFLD = SS+NASH combined) whether there is an association between hepatic n-3 PUFA content and gene expression. The third aim is to determine the intestinal microbiome (microbial composition and metagenome) in patients with SS or NASH and healthy controls.

DETAILED DESCRIPTION:
NASH is associated with obesity, diabetes and hyperlipidemia. Fat accumulation in the liver is likely due to variable degrees of disordered fatty-acid metabolism and insulin resistance (IR). Liver steatosis, especially polyunsaturated fatty acids (PUFA) in the liver, increases lipid peroxidation and is associated with a reduction in the antioxidant defense system. This oxidative stress can lead to increased production of pro-inflammatory cytokines (TNF-α, transforming growth factor-beta) contributing to the development of steatohepatitis and fibrosis.TNF-α - may further contribute to IR. In addition, changes in fatty acid composition within the liver may influence lipid metabolism and inflammation. In particular, n-3 PUFA have an effect on the insulin sensitivity, transcription of antioxidant genes, inflammatory response and production of reactive oxygen species. Differences might be seen on the gene expression level (mRNA) and also in epigenetic regulation (miRNA).

Microbiota composition might influence energy metabolism, and inflammatory tone and IR through increased endotoxemia and therefore could also play a role in the development of NAFLD.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients, age >18 y
* A liver biopsy with a diagnosis of SS or NASH OR No signs of steatosis, fibrosis or any other kind of liver disease on histology (minimal findings) OR For healthy control subjects, those with normal liver enzymes and normal liver imaging on ultrasound
* alcohol consumption (<20g of ethanol per day);
* absence of any other possible cause for liver dysfunction.

Exclusion criteria:

* any other liver disease apart from NAFLD
* anticipated need for liver transplantation in one year or complications of liver disease;
* any reasons contraindicating a liver biopsy (patients) or liver donation (healthy donors)
* chronic gastrointestinal diseases, previous gastrointestinal surgery modifying the anatomy, patients with diabetes requiring insulin.
* medications known to precipitate steatohepatitis (corticosteroids, high dose estrogens, methotrexate, amiodarone, spironolactone, sulfasalazine, perhexiline maleate, diethylamino- ethoxyhexestrol (DH), tamoxifen, diethylstilbestrol, naproxen or oxacillin) or regular intake of non-steroidal anti-inflammatory drugs (except for low dose aspirin), use of ursodeoxycholic acid or any experimental drug in the 6 months prior to entry.
* regular intake of prebiotics, probiotics, antibiotics, or laxatives; in the 3 months prior to study entry
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy living liver donors from the Multiorgan transplant program at the University Health Network Patients with nonalcoholic fatty liver disease (SS or NASH on liver biopsy) or patients with elevated liver enzymes but no significant findings on liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2003-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Hepatic fatty acid composition in total lipids in liver biopsy | Baseline
  Gas chromatography
Hepatic gene expression | Baseline
  mRNA by microarray
Intestinal microbiota composition | Baseline
  Illumina 16S technology

SECONDARY OUTCOMES:
Lipid peroxides in the liver | Baseline
  Test kit
Hepatic liver antioxidant power | Baseline
  Test kit
Hepatic microRNA expression in the liver | Baseline
  NanoString
Intestinal microbiota - specific organisms and groups | Baseline
  Quantitative real-time polymerase chain reaction
Intestinal microbiome on a genetic level | Baseline
  Illumina sequencing technology
Short-chain fatty acids in stool | Baseline
  Gas chromatography
Plasma endotoxin | Baseline
  Limulus assay

OTHER OUTCOMES:
Hepatic phospholipid composition | Baseline
  Gas chromatography
Red blood cell fatty acid and phospholipid composition | Baseline
  Gas chromatography
Plasma fatty acid composition | Baseline
  Gas chromatography
Plasma lipid peroxides | Baseline
  Test kit
Plasma antioxidant vitamins | Baseline
  Vitamin C colorimetric, alpha- and gamma-tocopherol and beta-carotene by high-performance liquid chromatography
Serum antioxidant power | Baseline
  Test kit
TNF-alpha in the liver | Baseline
  Enzyme linked immunosorbent assay
Immunohistochemistry | Baseline
  Staining for malondialdehyde, alpha-smooth muscle actin, transforming growth factor beta
Free choline in serum | Baseline
  liquid chromatography/electrospray ionization-isotope dilution mass spectrometry (LC/ESI-IDMS)
Bacterial DNA in plasma | Baseline
  Quantitative polymerase chain reaction for bacterial 16S rDNA
Insulin resistance | Baseline
  Fasting glucose and insulin to calculate insulin resistance (HOMA-IR), C-peptide, hemoglobin A1c, all by standard laboratory methods
Plasma ethanol | Baseline
  standard laboratory measurement
Anthropometry | Baseline
  Weight, height, skinfolds, bioelectrical impedance analysis
Food intake | Baseline
  7-day food records
Physical activity | Baseline
  7 day activity logs
Factors influencing intestinal microbiota | Baseline
  Environmental questionnaire
Liver function tests | Baseline
  Alanine transaminase, aspartate transaminase, alkaline phosphatase, standard laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD,FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Schwenger KJ, Allard JP. Clinical approaches to non-alcoholic fatty liver disease. World J Gastroenterol. 2014 Feb 21;20(7):1712-23. doi: 10.3748/wjg.v20.i7.1712. PMID 24587650
- [Background] Monteiro J, Leslie M, Moghadasian MH, Arendt BM, Allard JP, Ma DW. The role of n - 6 and n - 3 polyunsaturated fatty acids in the manifestation of the metabolic syndrome in cardiovascular disease and non-alcoholic fatty liver disease. Food Funct. 2014 Mar;5(3):426-35. doi: 10.1039/c3fo60551e. PMID 24496399
- [Background] Mouzaki M, Allard JP. The role of nutrients in the development, progression, and treatment of nonalcoholic fatty liver disease. J Clin Gastroenterol. 2012 Jul;46(6):457-67. doi: 10.1097/MCG.0b013e31824cf51e. PMID 22469640
- [Background] Mouzaki M, Allard J. Non-alcoholic steatohepatitis: the therapeutic challenge of a global epidemic. Ann Gastroenterol. 2012;25(3):207-217. PMID 24713803
- [Result] Da Silva HE, Arendt BM, Noureldin SA, Therapondos G, Guindi M, Allard JP. A cross-sectional study assessing dietary intake and physical activity in Canadian patients with nonalcoholic fatty liver disease vs healthy controls. J Acad Nutr Diet. 2014 Aug;114(8):1181-94. doi: 10.1016/j.jand.2014.01.009. Epub 2014 Mar 14. PMID 24631112
- [Result] Arendt BM, Ma DW, Simons B, Noureldin SA, Therapondos G, Guindi M, Sherman M, Allard JP. Nonalcoholic fatty liver disease is associated with lower hepatic and erythrocyte ratios of phosphatidylcholine to phosphatidylethanolamine. Appl Physiol Nutr Metab. 2013 Mar;38(3):334-40. doi: 10.1139/apnm-2012-0261. Epub 2012 Oct 15. PMID 23537027
- [Result] Mouzaki M, Comelli EM, Arendt BM, Bonengel J, Fung SK, Fischer SE, McGilvray ID, Allard JP. Intestinal microbiota in patients with nonalcoholic fatty liver disease. Hepatology. 2013 Jul;58(1):120-7. doi: 10.1002/hep.26319. Epub 2013 May 14. PMID 23401313
- [Result] Allard JP, Aghdassi E, Mohammed S, Raman M, Avand G, Arendt BM, Jalali P, Kandasamy T, Prayitno N, Sherman M, Guindi M, Ma DW, Heathcote JE. Nutritional assessment and hepatic fatty acid composition in non-alcoholic fatty liver disease (NAFLD): a cross-sectional study. J Hepatol. 2008 Feb;48(2):300-7. doi: 10.1016/j.jhep.2007.09.009. Epub 2007 Nov 20. PMID 18086506
- [Result] Arendt BM, Comelli EM, Ma DW, Lou W, Teterina A, Kim T, Fung SK, Wong DK, McGilvray I, Fischer SE, Allard JP. Altered hepatic gene expression in nonalcoholic fatty liver disease is associated with lower hepatic n-3 and n-6 polyunsaturated fatty acids. Hepatology. 2015 May;61(5):1565-78. doi: 10.1002/hep.27695. Epub 2015 Feb 27. PMID 25581263
- [Derived] Pasini E, Baciu C, Angeli M, Arendt B, Pellegrina D, Reimand J, Patel K, Tomlinson G, Mazhab-Jafari MT, Kotra LP, Fischer S, Allard JP, Humar A, Bhat M. Acyl-CoA Thioesterase 1 Contributes to Transition of Steatosis to Metabolic-Associated Steatohepatitis. Int J Hepatol. 2024 Jul 11;2024:5560676. doi: 10.1155/2024/5560676. eCollection 2024. PMID 39624175
- [Derived] Schwenger KJP, Sharma D, Ghorbani Y, Xu W, Lou W, Comelli EM, Fischer SE, Jackson TD, Okrainec A, Allard JP. Links between gut microbiome, metabolome, clinical variables and non-alcoholic fatty liver disease severity in bariatric patients. Liver Int. 2024 May;44(5):1176-1188. doi: 10.1111/liv.15864. Epub 2024 Feb 14. PMID 38353022
- [Derived] Pettinelli P, Arendt BM, Schwenger KJP, Sivaraj S, Bhat M, Comelli EM, Lou W, Allard JP. Relationship Between Hepatic Gene Expression, Intestinal Microbiota, and Inferred Functional Metagenomic Analysis in NAFLD. Clin Transl Gastroenterol. 2022 Jul 1;13(7):e00466. doi: 10.14309/ctg.0000000000000466. Epub 2022 Feb 10. PMID 35166723